CLINICAL TRIAL: NCT05934253
Title: The Effects of Low Viscosity Chloroprocaine Ophthalmic Gel 3% on the Bactericidal Action of Povidone-Iodine: A Comparison vs Tetracaine 0.5% Solution.
Brief Title: The Effects of Low Viscosity Chloroprocaine Ophthalmic Gel 3% on the Bactericidal Action of Povidone-Iodine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Harrow Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IZ-4-001
Record Dates: First submitted 2023-06-09; First posted 2023-07-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2023-09

CONDITIONS: Antiseptic; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chloroprocaine ophthalmic gel 3% (Experimental): FDA approved topical ophthalmic anesthetic applied 3 drops to the ocular surface before the planned procedure.
  Interventions: Drug: Chloroprocaine ophthalmic gel 3%
- Tetracaine ophthalmic solution 0.5% (Active Comparator): FDA approved topical ophthalmic anesthetic applied 3 drops to the ocular surface before the planned procedure.
  Interventions: Drug: Chloroprocaine ophthalmic gel 3%

INTERVENTIONS:
Drug: Chloroprocaine ophthalmic gel 3% — FDA approved topical ophthalmic anesthetic applied 3 drops to the ocular surface before the planned procedure.
  Other Names: Iheezo

SUMMARY:
To evaluate if Iheezo's (chloroprocaine 3%) gel vehicle acts as a barrier on the ocular surface, potentially blocking the bactericidal action of povidone-iodine.

DETAILED DESCRIPTION:
Choice in vehicle plays a large role in drug delivery with topical ophthalmic medications. One strategy to increase efficacy is by increasing the ocular surface contact time of a drug on the eye, primarily by increasing the viscosity of the vehicle. However, studies have demonstrated that high viscosity topical medications act as a barrier to subsequent drops. This poses a serious issue in pre-operative prophylaxis, as high viscosity vehicles may block the bactericidal action of povidone-iodine. This has been supported by in vitro studies of Akten (lidocaine 3.5%) gel.

Akten gel has a viscosity between 4000-9000 cps. Iheezo has a viscosity between 1200-2000 cps. Generic tetracaine 0.5% has a viscosity between 15-25cps. Healthy human tears have a viscosity of around 8 cps. For a vehicle to not act as a barrier to subsequent drops, it is believed that the viscosity should be close to human tears.

This study theorizes that Iheezo's lower viscosity will not act as a barrier to the bactericidal action of Povidone-iodine 5%.

This is a single site, prospective, randomized, patient masked, open-label study evaluating the effects of Iheezo (chloroprocaine HCl ophthalmic gel 3%) and how it may interact with povidone-iodine compared to tetracaine 0.5% ophthalmic solution. Consented patients will have their eyes randomized, one receiving Iheezo and the other tetracaine 0.5% ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients over age 18.
* Able to comprehend and sign a statement of informed consent.

Exclusion Criteria:

* Ocular surgery (e.g., intraocular, oculoplastic, corneal, or refractive surgical procedure) performed within the last 3 months or at any time that in the investigator's clinical judgment if it would interfere with the outcome measures of this study.
* Clinically significant ocular trauma.
* Diagnosis of lagophthalmos, or other severe eyelid abnormalities (entropion, ectropion, tumor, edema, blepharospasm, severe trichiasis, severe ptosis.)
* Active ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis) at the discretion of the investigator.
* Active ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection or the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye).
* Ocular infection within the last 3 months.
* Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis.
* Patients who are under age 18, pregnant or breastfeeding, or who may become pregnant during participation in the study.
* Monocular patients.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Change in colony forming units | Baseline and 5 minutes after baseline.
  Comparison of results from Bacterial Culture Swabs before and after application of drug and povidone-iodine. First bacterial culture at initiation. Study medication applied after culture. Povidone-iodine applied two minutes after. Second bacterial culture three minutes after.

CONTACTS AND LOCATIONS:
Locations (1):
- Brandon Eye Associates, Brandon, Florida, United States

IPD SHARING:
Plan to Share IPD: No